CLINICAL TRIAL: NCT00277368
Title: Headache in Epileptic Patients
Brief Title: A Study of the Prevalence of Headache in Epileptic Patients
Status: Completed | Type: Observational
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Clinical Research Director, Janssen Korea, Ltd., Korea
Other Study IDs: CR003613
Record Dates: First submitted 2006-01-13; First posted 2006-01-16 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Epilepsy
Keywords: Epilepsy; Headache; Seizure
MeSH Terms: conditions — Epilepsy; Headache; Seizures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- 001
  Interventions: Other: A structured questionnaire for seizure-related headache

INTERVENTIONS:
Other: A structured questionnaire for seizure-related headache — A structured questionnaire for seizure-related headache

SUMMARY:
The purpose of this study is to investigate the prevalence, characteristics and classification of headaches in epileptic patients.

DETAILED DESCRIPTION:
Headache is often ignored as a symptom of epileptic seizures. The purpose of this survey is to investigate the prevalence, characteristics and classification of seizure-associated headaches and non-seizure-associated headaches in epileptic patients in Korea, according the criteria of the International Headache Society 2004. In this survey, 577 consecutive patients with a recent diagnosis of epilepsy are interviewed by questionnaire about headaches associated with epileptic seizures. It involves questions about headache in general, localization, severity, duration and frequency, as well as headache associated with seizures, and about patient's family history. This Observational study does not involve the administration of any drugs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a recent diagnosis epilepsy
* Able to describe their symptoms by themselves
* Have had at least 2 episodes of seizures during the previous year
* Have had at least 1 headache during the previous year

Exclusion Criteria:

* Well-controlled epileptic patients taking anti-epileptic medications

Ages: 13 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a recent diagnosis epilepsy; able to describe their symptoms by themselves; have had at least 2 episodes of seizures during the previous year; have had at least 1 headache during the previous year.
Sampling Method: Non-Probability Sample
Enrollment: 719 (Actual)
Dates: Start 2005-07; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Rate of seizure-related headache among epilepsy patients and its classification | At first visit (This study is cross-sectional)

SECONDARY OUTCOMES:
The pain intensity of seizure-related headache | At 1st visit
The frequency of seizure-related headache | At 1st visit

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd. Clinical Trial, Study Director — Janssen Korea, Ltd.